CLINICAL TRIAL: NCT05442619
Title: Developing a Portable Therapeutic Baby Nest for Newborns and Evaluation of the Effect on Comfort and Pain Levels During Venous Blood Collection
Brief Title: Developing a Portable Therapeutic Baby Nest for Newborns and Evaluation During Venous Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, AYLİN ARIKAN, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 56786525-050.04.04/385491
Record Dates: First submitted 2022-06-23; First posted 2022-07-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Pain; Newborn; Comfort
Keywords: light; noise; baby nest; pediatric emergency
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Control Group Portable Therapeutic Baby Nest Using Group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portable therapeutic baby nest group (Experimental): Blood will be drawn from newborns using the portable therapeutic baby nest.
  Interventions: Procedure: Venous blood collection
- Control group (Active Comparator): Blood collection from newborns will be done according to the clinical routine.
  Interventions: Procedure: Venous blood collection

INTERVENTIONS:
Procedure: Venous blood collection — Venous blood will be drawn from newborns.

SUMMARY:
The neonatal period covers the first 28 days after birth. Newborns may experience problems such as jaundice, restlessness, nasal congestion, respiratory distress, and vomiting in this process, and for these reasons, children are brought to the emergency services. From the moment they enter the emergency service, they are exposed to sensory stimuli in the form of bright lights, loud and unusual sounds, and new tactile experiences. This creates an uncomfortable and stressful experience for them. At the same time, performing invasive procedural interventions in an environment where stimuli are intense causes pain. Newborns give physiological, behavioral and metabolic responses depending on the pain and stress they experience. Persistent exposure to these interventions and lack of appropriate approaches may lead to deterioration in pain perceptions and neuroendocrine stress responses, and permanent neurological and behavioral problems may develop over time. For this reason, pain in newborns and the problems caused by stress should be known, appropriate pain relief methods should be selected and comfort should be provided. However, pediatric emergency nurses who perform the procedural methods of newborns whose rates of admission to pediatric emergency services are reported as 2-3% may not have sufficient experience in pain management in newborns. Pediatric emergency nurses need to be supported in order to increase their awareness of newborns and to continue their pain management. While it has been reported in the literature that there are non-pharmacological methods including individualized developmental care practices in the procedural pain management of newborns; there are no studies aimed at reducing their pain, preventing their exposure to environmental factors and ensuring their comfort during painful procedures in pediatric emergency departments. In this context, it is planned to use a portable therapeutic baby nest in the pediatric emergency department, where newborns will feel safe and maintain their flexion posture during the venous blood sampling, as well as be protected from noise and light, thereby reducing the pain caused by the procedural method and providing comfort, and a randomized controlled experimental study.

DETAILED DESCRIPTION:
The neonatal period covers the first 28 days after birth. During this period, newborns may experience problems such as jaundice, restlessness, nasal congestion, respiratory distress, and vomiting, and for these reasons, children can be brought to the emergency services. From the moment they enter the emergency room, they are exposed to sensory stimuli in the form of bright lights, loud and unusual sounds, and new tactile experiences. This creates an uncomfortable and stressful experience for them. At the same time, performing invasive procedural interventions in an environment where stimuli are intense causes pain. Newborns give physiological, behavioral and metabolic responses depending on the pain and stress they experience. Persistent exposure to these interventions and lack of appropriate approaches may lead to deterioration in pain perceptions and neuroendocrine stress responses, and permanent neurological and behavioral problems may develop over time. For this reason, pain in newborns and the problems caused by stress should be known, appropriate pain relief methods should be selected and comfort should be provided. However, pediatric emergency nurses who perform the procedural procedures of newborns whose rates of admission to pediatric emergency services are reported as 2-3% may not have sufficient experience in pain management. Pediatric emergency nurses need to be supported in order to increase their awareness of newborns and to continue their pain management. Although there is a large literature examining the effects of individualized developmental care practices in painful invasive procedural procedures for newborns, there are no studies examining the effects of these practices in painful invasive procedural procedures in pediatric emergencies. In this context, there is a need for an environment in which invasive procedural procedures specific to them are carried out in pediatric emergency services for newborns with the highest sensitivity to environmental factors and susceptibility to infections. In this study, newborns will feel safe, protect their flexion posture, and be protected from noise and light during the venous blood collection procedure, which is unique and cost-effective in terms of its applicability in each pediatric emergency department, thus reducing the pain caused by the procedural procedure and providing comfort. It is aimed to develop and evaluate the effectiveness of the portable therapeutic baby nursery. With these aspects, it is the first study in the literature to be conducted in the pediatric emergency department and will be carried out in two stages. In the first stage of the study, a portable therapeutic baby nursery will be developed, and in the second stage, its effectiveness during venous blood collection will be evaluated. Nest is an environment specific to newborns in the medical field; thanks to its design; It helps newborns to reduce the light and sound that they will be exposed to in a noisy and high light environment such as a pediatric emergency, to provide comfort and reduce pain by therapeutic touch and maintaining their therapeutic position, at the same time to protect body temperature by preventing contact with cold material such as linoleum on the stretcher and over the stretcher. will contribute to the prevention of exposure to any infectious agent. Thanks to this new and field-specific application, information about the individualized developmental care practices of newborns in the pediatric emergency service will be provided to the literature.

ELIGIBILITY:
Inclusion Criteria:

* 37-42 weeks of gestation,
* Birth weight between 2500-4000 g,
* Being less than 28 postnatal days,
* The family can speak and understand Turkish,
* Newborns with written and verbal informed consent from their families

Exclusion Criteria:

* Having an analgesic intake 4 hours before, which may affect their comfort and behavior
* Presence of congenital anomaly,
* Having respiratory distress,
* Newborns with clinically unstable (vital and physical examination findings)
* Newborns with suspected or diagnosed Covid 19
* Newborns with vision and hearing problems
* Inability to perform blood collection at once
* Newborns have a history of hospitalization

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Prosedural Pain | In each infant, the level of pain will be evaluated in an average of 6 minutes.
  "The Neonatal-Infant Pain (NIPS) Scale" will be used to measure the pain levels of newborns during the blood collection.
  Neonatal Infant Pain Scale (NIPS): The Neonatal Infant Pain Scale (NIPS), developed by Lawrence et al. (1993), is a behavioral scale and can be used with both full-term and preterm infants. In NIPS, five behavioral indicators (facial expression, cry, arms, legs, and state of arousal) and one physiological parameter (breathing pattern) are assessed. The total pain score ranges between 0 and 7 with 0-2 points indicating mild to no pain, 3-4 indicating mild to moderate pain, and greater than 4 indicating severe pain (Lawrence et al., 1993). The scale was adapted to Turkish. Cronbach alpha internal consistency coefficient was found between 0.83 and 0.86 (Akdovan et al., 1999).
Comfort | In each infant, the level of comfort will be evaluated in an average of 6 minutes.
  "COMFORTneo Scale" will be used to measure the comfort levels of newborns during the blood collection.
  COMFORTneo Scale: The COMFORTneo scale is used to assess the comfort levels of infants. This scale is a Likert-type scale consisting of seven parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tonus. The lowest score on the scale is 6 and the highest is 30. If the total score of the scale is between 14 and 30, the infant has pain or distress, is uncomfortable, and needs intervention to provide comfort. The validity and reliability study of the Turkish version of the scale was conducted. Cronbach's alpha coefficient of the scale was 0.82-0.92 (Kahraman et al., 2014).
Physiological parameters- Pulse rate | In each infant, the level of physiologic parameters will be evaluated in an average of 6 minutes.
  Pulse oximeter will be used to record data about pulse rate (beats/minute).Pulse rate will be recorded under the titles of 2 minute before the procedure, during the procedure (during the blood collection), and 2 minutes after the procedure; Total duration (of the procedure) will be recorded in seconds.
Physiological parameters- Oxygen saturation | In each infant, the level of physiologic parameters will be evaluated in an average of 6 minutes
  Pulse oximeter will be used to record data about oxygen saturation (SpO2).Oxygen saturation will be recorded under the titles of 2 minute before the procedure, during the procedure (during the blood collection), and 2 minutes after the procedure; Total duration (of the procedure) will be recorded in seconds.
Physiological parameters-Respiration rate | In each infant, the level of physiologic parameters will be evaluated in an average of 6 minutes
  A smartphone stopwatch will be used to measure respiratory rate (breaths/minute). Respiratory rate will be recorded under the titles of 2 minute before the procedure, during the procedure (during the blood collection), and 2 minutes after the procedure; Total duration (of the procedure) will be recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sami Ulus Maternity and Child Health and Diseases Training and Research Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Derived] Arikan A, Esenay FI. Effect of a portable therapeutic baby nest designed for neonates on physiological parameters, comfort and pain levels during venous blood sampling: a randomised controlled trial. Emerg Med J. 2025 Oct 20;42(11):705-711. doi: 10.1136/emermed-2024-214660. PMID 40634119